CLINICAL TRIAL: NCT05159492
Title: Ground-Breaking Electroporation-based Intervention for PAROXysmal Atrial Fibrillation Treatment (BEAT PAROX-AF)
Acronym: BEAT PAROX-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2021/03
Record Dates: First submitted 2021-12-01; First posted 2021-12-16 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Cardiac Arrhythmia; Pulmonary vein Isolation; Catheter Ablation; RF Ablation; Pulsed Field Energy
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Open-label randomised controlled trial, in two parallel groups with a 1:1 allocation ratio
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PEF Arm (Experimental): PEF is a non-thermal ablation modality using extremely short high voltage pulses to induce cell death, with tissue selectivity, cardiomyocytes being much more sensitive to this energy than Phrenic nerve or Esophageal cells. Energy (2000 V) will be delivered 8 times per vein with 2 different catheter configurations and rotations
  Interventions: Device: PVI using PEF
- Pulmonary vein isolation using Contact Force RF (Active Comparator): The PVI strategy using RF is very standard. The CARTO© platform will be used, with a contact force catheter (SmartTouch), aiming at an ablation index value of 300 to 400 on the posterior wall, and at least 500 on the anterior wall. Power will be limited to 35/45 W, with a distance between consecutive deliveries of 6 mm or less (CLOSE protocol).
  Interventions: Device: PVI using CFRF

INTERVENTIONS:
Device: PVI using PEF — PVI using PEF
  Arms: PEF Arm
Device: PVI using CFRF — PVI using CFRF
  Arms: Pulmonary vein isolation using Contact Force RF

SUMMARY:
BEAT AF is a randomized controlled trial aiming to demonstrate that pulsed field energy is faster, more effective and safer (tissue selectivity) than RF for paroxysmal AF ablation

DETAILED DESCRIPTION:
Atrial fibrillation (AF), the most common arrhythmia, accounts for 1/3rd of Cardiovascular expenses, with over 10 millions affected in Europe. In addition to significant impact on quality of life, AF exposes patients to stroke, heart failure, dementia and death. AF is the most commonly ablated arrhythmia. The Pulmonary Vein Isolation (PVI) is the cornerstone of AF ablation, preventing recurrences, especially in patients with paroxysmal AF. Catheter ablation of AF uses either radiofrequency (RF) or cryothermal (cryo) energy. Common to these thermal energy sources is their reliance on time-dependent conductive heating/cooling and the fact that these modalities ablate all tissue types indiscriminately. The ablation procedure remains long, requires skills and expertise, and has a limited success rate, mostly because of non-durable lesions after PVI implying frequent redo procedures. And these energies are associated with rare but severe complications due to their thermal nature. The goal of BEAT AF is to disrupt AF ablation by achieving durable PVI with permanent, coalescent and transmural ablation lesions using Pulsed Electric Field (PEF) energy. PEF is non-thermal and creates nanoscale pores in cell membranes. Cardiac cells are highly sensitive to PEF unlike phrenic and oesophageal cells. BEAT AF aims to demonstrate that PEF ablation is faster, more effective and safer (tissue selectivity) than RF ablation to treat paroxysmal AF. For this purpose, a randomized clinical trial will be conducted to provide first comparative evidence of the superiority of PEF over RF on the rate of 1-year recurrence for paroxysmal AF. The BEAT AF consortium gathers 9 European renowned clinical centres (France, Czech Republic, Germany, Austria, Belgium) to contribute to decrease the huge burden of AF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with drug-resistant symptomatic PAF meeting all the following criteria:

   1. Paroxysmal: AF that terminates spontaneously or with intervention within 7 days of onset.
   2. Frequency:

   i. Physician documentation of recurrent PAF (two or more episodes) within 6 months, AND ii. At least one (1) documented episode by a recording such as ECG, Event Monitor, Holter monitor or telemetry strip within 12 months of enrolment.

   c. Drug failed: Failed AAD treatment, meaning therapeutic failure of at least one (1) AAD (Class I to IV) for efficacy and / or intolerance.
2. Patients who are ≥ 18 and ≤ 75 years of age on the day of enrollment.
3. Patient who are willing and capable of:

   1. Providing informed consent to undergo study procedures AND
   2. Participating in all examinations and follow-up visits and tests associated with this clinical study.
   3. Patient having a smart phone compatible with the Event Monitor device.
4. Effective contraception for women of childbearing potential.
5. Effective oral anticoagulation >3 weeks prior to planned ablation procedure
6. Patient affiliated to or beneficiary of national health security scheme for French participants.

Exclusion Criteria:

* 1. AF that is any of the following:

  1. Persistent (both early and longstanding) by diagnosis or continuous duration > 7 days
  2. Secondary to electrolyte imbalance, thyroid disease, alcohol or other reversible / non-cardiac causes 2. Any of the following atrial conditions:

  <!-- -->

  1. Left atrial anteroposterior diameter ≥ 5.5 cm (by MRI, CT or TTE)
  2. Any prior atrial endocardial or epicardial ablation procedure, other than right sided cavotricuspid isthmus ablation or for right sided SVT
  3. Any prior atrial surgery
  4. Intra-atrial septal patch or interatrial shunt
  5. Atrial myxoma
  6. Current LA thrombus
  7. LA appendage closure, device or occlusion, past or anticipated
  8. Any PV abnormality, stenosis or stenting (common and middle PVs are admissible) 3. At any time, one (1) or more of the following cardiovascular procedures, implants or conditions:

  a. Sustained ventricular tachycardia or any ventricular fibrillation b. Hemodynamically significant valvular disease: i. Valvular disease that is symptomatic ii. Valvular disease causing or exacerbating congestive heart failure iii. Aortic stenosis: if already characterized, valve area < 1.5cm or gradient > 20 mm Hg iv. Mitral stenosis: if already characterized, valve area < 1.5cm or gradient > 5 mm Hg v. Aortic or mitral regurgitation associated with abnormal LV function or hemodynamic measurements c. Hypertrophic cardiomyopathy d. Any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty e. Pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices f. Any inferior vena cava (IVC) filter, known inability to obtain vascular access or other contraindication to femoral access g. History of rheumatic fever h. History of congenital heart disease with any residual anatomic or conduction abnormality 4. Any of the following procedures, implants or conditions:

  a. At baseline: i. New York Heart Association (NYHA) Class III/IV ii. Left ventricular ejection fraction (LVEF) < 40% iii. Symptomatic hypotension iv. Uncontrolled hypertension (SBP > 160 mmHg or DBP > 95 mmHg on two BP measurements at baseline assessment) v. Symptomatic resting bradycardia vi. Implantable loop recorder or insertable cardiac monitor, b. Within the 3 months preceding the Consent Date: i. Myocardial infarction ii. Unstable angina iii. Percutaneous coronary intervention iv. Heart failure hospitalization v. Pericarditis or symptomatic pericardial effusion vi. Gastrointestinal bleeding c. Within the 6 months preceding the Consent Date: i. Heart surgery ii. Stroke, TIA or intracranial bleeding iii. Any thromboembolic event iv. Carotid stenting or endarterectomy 5. Diagnosed disorder of blood clotting or bleeding diathesis 6. Contraindication to, or unwillingness to use, systemic anticoagulation 7. Contraindication to both CT and MRI 8. Sensitivity to contrast media not controllable by premedication 9. Women of childbearing potential who are pregnant, lactating, not using medical birth control or who are planning to become pregnant during the anticipated study period 10. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation, including but not limited to:
  1. Body Mass Index (BMI) > 40.0
  2. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
  3. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
  4. Renal insufficiency with an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
  5. Active malignancy or history of treated malignancy within 24 months of enrollment (other than cutaneous basal cell or squamous cell carcinoma)
  6. Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
  7. Active systemic infection
  8. COVID-19 disease
  9. Current confirmed, active COVID-19 disease ii. Current positive test for SARS-CoV-2 iii. Confirmed COVID-19 disease not clinically resolved at least 3 months prior to the Consent Date.

  i. Other uncontrolled medical conditions that may modify device effect or increase risk, including uncontrolled diabetes mellitus (HgbA1c > 8.0% if test result already obtained), untreated obstructive sleep apnea or active alcohol abuse j. Predicted life expectancy less than one (1) year 11. Clinically significant psychological condition that in the Investigator's opinion would prohibit the subject's ability to meet the protocol requirements/ Patient under legal protection 12. Current or anticipated enrollment in any other clinical study. 13. Employees / family members of:
  1. FARAPULSE or any of its affiliates or contractors
  2. The Investigator, sub-Investigators, or their medical office or practice, or healthcare organizations at which study procedures may be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
proportion of subjects experiencing 1-year single-procedure clinical success | 1 year
  The Primary Efficacy Endpoint is the proportion of subjects experiencing 1-year single-procedure clinical success, defined as (2017 HRS consensus statement):
  1. Successful index AF ablation
  2. Absence of atrial arrhythmia recurrence on any type of recording (≥ 30 sec by TTM (event monitor), Holters, 12-lead ECGs, rhythm strip or other diagnostic ECG documentation),
  3. Absence of use of class I or III AAD (except for non-atrial arrhythmia)
  4. Absence of redo ablation (except for typical flutter), in the 12 months following the index ablation procedure (including a blanking period of 60 days following the index ablation procedure).

SECONDARY OUTCOMES:
proportion of subjects with 1-year multiple-procedures success | 1 year
  proportion of subjects with 1-year multiple-procedures success defined as the following up to 12 months following the index ablation procedure:
  1. Absence of atrial arrhythmia recurrence on any type of recording ((≥ 30 sec by TTM (event monitor), Holters, 12-lead ECGs, rhythm strip or other diagnostic ECG documentation),
  2. Absence of use of class I or III AAD (except for non-atrial arrhythmia)
health-related quality of life: | 6 months, 1 year
  Health-related quality of life will be evaluated using the SF-12 questionnaire. The SF-12 includes 8 concepts commonly represented in health surveys: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health. Results are expressed in terms of two meta-scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). High score indicates better functioning
AF-specific quality of life | 6 months, 1 year
  Improvement in AF-specific quality of life will be assessed using QualiTy-of-life (AFEQT) questionnaire. Scores range from 0 to 100. A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered)
Death | 7 days, 1 year
  Proportion of participants with death
Stroke | 7 days, 1 year
  Proportion of participants with
Embolic events from arrhythmia, | 1 year
  Proportion of participants with embolic events from arrhythmia
Myocardial infarction | 7 days
  Proportion of participants with Myocardial infarction
Persistent diaphragmatic paralysis | 7 days
  Proportion of participants with Persistent diaphragmatic paralysis
Transient ischemic attack (TIA) | 7 days
  Proportion of participants with Transient ischemic attack (TIA)
Peripheral or organ thromboembolism | 7 days
  Proportion of participants with Peripheral or organ thromboembolism
Cardiac Tamponade / Perforation | 7 days
  Proportion of participants with Cardiac Tamponade / Perforation
Pericarditis | 7 days
  Proportion of participants with Pericarditis
Hospitalisation | 7 days
  Proportion of participants with Hospitalisation (initial or prolonged), excluding hospitalisation solely due to arrhythmia recurrence
Heart block | 7 days
  Proportion of participants with Heart block
Vascular access complications | 7 days
  Proportion of participants with Vascular access complications
Pulmonary vein stenosis (PVS) | 1 year
  Proportion of participants with Pulmonary vein stenosis (PVS)
Atrio-oesophageal fistula | 1 year
  Proportion of participants with Atrio-oesophageal fistula
Total ablation procedure duration | Baseline
  Index Ablation Procedure parameters: Total ablation procedure duration (in minutes), skin to skin
Left atrial (LA) dwell time during ablation procedure | Baseline
  Index Ablation Procedure parameters: Left atrial (LA) dwell time, defined as the time (in minutes) transpiring from catheter entry to exit from the LA
Total fluoroscopy time during ablation procedure | Baseline
  Index Ablation Procedure parameters: Total fluoroscopy time (in minutes), skin-to-skin
PV diameter | 2 months
  Change in mean PV diameter 2 months
Incidence of acute vagal response during PVI | Baseline
  Incidence of acute vagal response during PVI
mean heart rate | 1 year
  Change in mean heart rate
heart rate variability | 1 year
  Change in heart rate variability

CONTACTS AND LOCATIONS:
Locations (9):
- Medical University of Graz, Graz, Austria
- AZ Sint-Jan Brugge-Oostende, Bruges, Belgium
- Czechia (2):
  - Homolka Hospital, Prague
  - Institute for Clinical and Experimental Medicine, Prague
- France (3):
  - CHU Bordeaux, Pessac
  - CHU Toulouse, Toulouse
  - Clinique Pasteur, Toulouse, Toulouse
- Germany (2):
  - Cardiovascular Center Bad Neustadt, Bad Neustadt an der Saale
  - Deutsches Herzzentrum München, Munich

IPD SHARING:
Plan to Share IPD: Undecided